CLINICAL TRIAL: NCT05685810
Title: Genetic and Clinical Determinants of Cardiovascular Disease, Diabetes, Kidney Disease and Obesity in People of African Ancestry With HIV
Brief Title: Genetic Determinants of Kidney Disease in People of African Ancestry With HIV
Acronym: GEN-AFRICA
Status: Active, not recruiting | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); Lewisham and Greenwich NHS Trust (Other Government); Royal Free Hospital NHS Foundation Trust (Other); Central and North West London NHS Foundation Trust (Other); Barts & The London NHS Trust (Other); Chelsea and Westminster NHS Foundation Trust (Other); Imperial College Healthcare NHS Trust (Other); North Middlesex University Hospital NHS Trust (Other Government); Brighton and Sussex University Hospitals NHS Trust (Other); The Leeds Teaching Hospitals NHS Trust (Other); Manchester University NHS Foundation Trust (Other Government); Newcastle-upon-Tyne Hospitals NHS Trust (Other); South Tees Hospitals NHS Foundation Trust (Other); Africa Advocacy Foundation (Unknown); Vanderbilt University (Other); University of Cape Town (Other); University of Pennsylvania (Other); Medical Research Council (Other Government); British HIV Association (Unknown); Gilead Sciences (Industry); St George's Healthcare NHS Trust (Other); Guy's & St Thomas' Charity (Other)
Responsible Party: Sponsor
Other Study IDs: 239895
Record Dates: First submitted 2023-01-03; First posted 2023-01-17 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-02

CONDITIONS: HIV Nephropathy; Kidney Injury; Kidney Diseases; Diabetes Mellitus; Obesity; Cardiovascular Diseases; Genetic Predisposition to Disease
MeSH Terms: conditions — AIDS-Associated Nephropathy; Kidney Diseases; Diabetes Mellitus; Obesity; Cardiovascular Diseases; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — DNA (from PBMC), urine, serum, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Black ethnicity is a major risk factor for chronic kidney disease [CKD] in people with HIV infection, suggesting that genetic factors are an important determinant of kidney disease progression in this population. The Gen-Africa study was established in 2018 to allow the study of genetic and clinical risk factors for CKD in people with HIV in the UK. Just over 3000 people across 15 sites were enrolled between May 2018 and January 2020. Demographic and clinical information was collected, and biological samples (buffy coats, plasma and urine) obtained. Cross-sectional analyses have revealed that participants of West-African ancestry are at higher risk of CKD and end-stage kidney disease [ESKD], and that genetic variants in the apolipoprotein L1 (APOL1) gene and sickle cell trait (SCT) are predictors of CKD and ESKD. The pathogenesis of APOL1- and SCT-associated CKD is incompletely understood, and additional, longitudinal data will be collected to improve understanding of the contribution of demographic, traditional CKD (diabetes, hypertension, obesity/metabolic syndrome, cardiovascular disease) and HIV (immuno-virological and hepatitis B/C co-infection status, antiretroviral medications) risk factors as well as additional genetic and epigenetic markers.

DETAILED DESCRIPTION:
At enrolment, just over 3,000 people of (self-identified) back ethnicity provided informed consent, a blood and urine sample, weight, height, and blood pressure measurements, and completed a short questionnaire about your health issues and lifestyle factors. HIV treatment history, including most recent and nadir CD4 count and HIV viral load, viral hepatitis status and kidney function measurements were recorded. Records for about 2,350 participants have been successfully linked to the United Kingdom Collaborative HIV Cohort (UK CHIC) which has collected data (demographics, clinical and laboratory parameters) on people with HIV since 1998 at selected clinics in the United Kingdom.

Several GEN-AFRICA sub-studies (CKD-AFRICA, Coronavirus disease (CoV)-AFRICA, Ob-AFRICA) have been conducted or are being planned. Each of these studies has received, or will be submitted for, regulatory approval. The studies have allowed or will allow collection of more detailed clinical information, additional biological samples, and/or through linkage with electronic clinical records, collection of longitudinal data on HIV (CD4, HIV viral load, AIDS-defining illnesses, and details of antiretroviral therapy), comorbidities (diabetes, hypertension, kidney disease, cardiovascular events), measurements such as blood pressure and weight, and results of blood tests including measures of kidney function performed as part of clinical monitoring.

Data collected as part of the GEN-AFRICA study / sub-studies are stored at King's College Hospital under their GEN-AFRICA/CKD-AFRICA/CoV-AFRICA/Ob-AFRICA study identifiers (ID). Samples collected as part of these protocols are labeled by study ID and stored in the James Black Building, King's College London, London, UK, in compliance with human tissue act (HTA) standards. Prof. Frank post is the custodian of the data and samples and will be responsible for ensuring all study activity is compliant with relevant data protection and other policies.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* Black ethnicity (self-identified)
* Informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Black people with HIV infection who received care at one of 15 HIV clinics in the United Kingdom.
Sampling Method: Non-Probability Sample
Enrollment: 3029 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Kidney disease | 2018-2030
  Incidence and predictors of end-stage kidney disease, chronic kidney disease, HIVAN, focal and segmental glomerulosclerosis (FSGS), tenofovir disoproxil fumarate (TDF)-associated kidney injury.

SECONDARY OUTCOMES:
Coronavirus disease (COVID-19) | 2020-2023
  Incidence and clinical and genetic determinants of COVID-19
Multi-morbidity | 2019-2023
  Clinical and social determinants of multi-morbidity
Weight change | 2013-2024
  Weight change in relation to antiretroviral exposures
Obesity | 2013-2024
  Incidence of obesity in relation to antiretroviral exposures
Dysglycaemia | 2019-2023
  Relationship between fasting blood glucose/HbA1c and waist circumference/BMI
Insulin resistance | 2019-2023
  Relationship between fasting blood glucose/HbA1c, insulin/C-peptide, and waist circumference/BMI

CONTACTS AND LOCATIONS:
Overall Officials: Frank A Post, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The database contains personal and sensitive information and is therefore not publicly available. Access to the study data and/or samples is governed by the National Health Service data access policy and those of King's College Hospital National Health System (NHS) Foundation Trust, the study sponsor. The Gen-AFRICA cohort is open to collaborations, and all requests from researchers who meet the criteria for access to fully anonymized patient level data will be considered.

REFERENCES:
- [Background] Ottaway Z, Campbell L, Fox J, Burns FM, Hamzah L, Schoeman S, Price D, Clarke A, Pett SL, Onyango D, Sabin C, Miller RF, Post FA; COVID-AFRICA study group. Post-acute sequelae of COVID-19 in people of Black ethnicities living with HIV in the United Kingdom. Int J STD AIDS. 2025 Jul;36(8):602-610. doi: 10.1177/09564624251334227. Epub 2025 Apr 14. PMID 40227084
- [Background] Moon Z, Campbell L, Ottaway Z, Fox J, Burns F, Hamzah L, Ustianowski A, Clarke A, Schoeman S, Sally D, Tariq S, Post FA, Horne R. Mapping Vaccination Mindsets among UK Residents of Black Ethnicities with HIV: Lessons from COVID-19. AIDS Behav. 2025 May;29(5):1516-1524. doi: 10.1007/s10461-025-04622-0. Epub 2025 Mar 10. PMID 40063203
- [Background] Ottaway Z, Onyango D, Kolodin V, Carter A, Horne R, Campbell L, Hamzah L, Post FA, Tariq S, Nicholls EJ. 'COVID impacted my life in so many ways': a qualitative study of the lived experiences of the COVID-19 pandemic among people of Black ethnicities living with HIV in England. Ethn Health. 2025 Feb;30(2):254-272. doi: 10.1080/13557858.2024.2429405. Epub 2024 Nov 26. PMID 39593273
- [Background] Kolodin V, Barbini B, Onyango D, Musomba R, Liu J, Hung RKY, Nikiphorou E, Campbell L, Post FA, Tariq S, Lempp H. Social determinants of health and long-term conditions in people of Black African and Black Caribbean ethnicity living with HIV in London: A qualitative study. Health Expect. 2024 Jun;27(3):e14055. doi: 10.1111/hex.14055. PMID 38666627
- [Background] Patel N, Post FA. Surveillance for hepatocellular carcinoma in people of African ancestry with HIV and Hepatitis B. Int J STD AIDS. 2022 Feb;33(2):202-204. doi: 10.1177/09564624211042828. Epub 2021 Sep 21. PMID 34546112
- [Background] Ko S, Dominguez-Dominguez L, Ottaway Z, Campbell L, Fox J, Burns F, Hamzah L, Ustianowski A, Clarke A, Kegg S, Schoeman S, Jones R, Pett SL, Hudson J, Post FA. Cardiovascular disease risk in people of African ancestry with HIV in the United Kingdom. HIV Med. 2024 Dec;25(12):1289-1297. doi: 10.1111/hiv.13706. Epub 2024 Aug 29. PMID 39209512
- [Background] Ottaway Z, Campbell L, Fox J, Burns F, Hamzah L, Kegg S, Rosenvinge M, Schoeman S, Price D, Jones R, Miller RF, Tariq S, Post FA. HIV outcomes during the COVID-19 pandemic in people of Black ethnicities living with HIV in England. HIV Med. 2024 Jul;25(7):885-892. doi: 10.1111/hiv.13640. Epub 2024 Mar 26. PMID 38529684
- [Background] Ottaway Z, Campbell L, Cechin LR, Patel N, Fox J, Burns F, Hamzah L, Kegg S, Rosenvinge M, Schoeman S, Price D, Jones R, Clarke A, Maan I, Ustianowski A, Onyango D, Tariq S, Miller RF, Post FA; COVID-AFRICA study group. Clinical epidemiology of COVID-19 in people of black ethnicity living with HIV in the UK. HIV Med. 2024 May;25(5):614-621. doi: 10.1111/hiv.13611. Epub 2024 Jan 11. PMID 38213094
- [Background] Dominguez-Dominguez L, Hamzah L, Fox J, Vincent RP, Post FA. Brief Report: Cystatin C Provides Substantially Higher Glomerular Filtration Rate Estimates Than Creatinine in a Subset of Black People With HIV on Current Antiretroviral Regimens. J Acquir Immune Defic Syndr. 2025 Feb 1;98(2):171-175. doi: 10.1097/QAI.0000000000003555. PMID 39791983
- [Background] Cechin L, Dominguez-Dominguez L, Campbell L, Hamzah L, Fox J, Vincent RP, Dimitriadis GK, Goff L, Post FA. Waist circumference and cardiometabolic parameters in people of African/Caribbean ancestry with HIV in South London (CKD-AFRICA study). Int J STD AIDS. 2024 Jun;35(7):521-526. doi: 10.1177/09564624241233036. Epub 2024 Feb 20. PMID 38377277
- [Background] Dominguez-Dominguez L, Campbell L, Barbini B, Fox J, Nikiphorou E, Goff L, Lempp H, Tariq S, Hamzah L, Post FA. Associations between social determinants of health and comorbidity and multimorbidity in people of black ethnicities with HIV. AIDS. 2024 May 1;38(6):835-846. doi: 10.1097/QAD.0000000000003848. Epub 2024 Feb 1. PMID 38265411
- [Background] Hung RKY, Costeira R, Chen J, Schlosser P, Grundner-Culemann F, Booth JW, Sharpe CC, Bramham K, Sun YV, Marconi VC, Teumer A, Winkler CA, Post FA, Bell JT. Epigenetic associations with kidney disease in individuals of African ancestry with APOL1 high-risk genotypes and HIV. Nephrol Dial Transplant. 2025 Apr 28;40(5):997-1006. doi: 10.1093/ndt/gfae237. PMID 39448372
- [Background] Hung RKY, Santana-Suarez B, Binns-Roemer E, Campbell L, Bramham K, Hamzah L, Fox J, Burns JE, Clarke A, Vincent R, Jones R, Price DA, Onyango D, Harber M, Hilton R, Booth JW, Sabin CA, Winkler CA, Post FA; GEN-AFRICA study group. The epidemiology of kidney disease in people of African ancestry with HIV in the UK. EClinicalMedicine. 2021 Jul 8;38:101006. doi: 10.1016/j.eclinm.2021.101006. eCollection 2021 Aug. PMID 34286237
- [Background] Hung RKY, Binns-Roemer E, Booth JW, Hilton R, Harber M, Santana-Suarez B, Campbell L, Fox J, Ustianowski A, Cosgrove C, Burns JE, Clarke A, Price DA, Chadwick D, Onyango D, Hamzah L, Bramham K, Sabin CA, Winkler CA, Post FA; GEN-AFRICA Study Group. Genetic Variants of APOL1 Are Major Determinants of Kidney Failure in People of African Ancestry With HIV. Kidney Int Rep. 2022 Jan 25;7(4):786-796. doi: 10.1016/j.ekir.2022.01.1054. eCollection 2022 Apr. PMID 35497797
- [Background] Hung RKY, Binns-Roemer E, Booth JW, Hilton R, Fox J, Burns F, Harber M, Ustianowski A, Hamzah L, Burns JE, Clarke A, Price DA, Kegg S, Onyango D, Santana-Suarez B, Campbell L, Bramham K, Sharpe CC, Sabin CA, Winkler CA, Post FA; GEN-AFRICA Study Group. Sickle Cell Trait and Kidney Disease in People of African Ancestry With HIV. Kidney Int Rep. 2021 Dec 13;7(3):465-473. doi: 10.1016/j.ekir.2021.12.007. eCollection 2022 Mar. PMID 35257059
- [Background] Hung RKY, Rosenberg KL, David V, Binns-Roemer E, Booth JW, Hilton R, Fox J, Burns F, Ustianowski A, Cosgrove C, Hamzah L, Burns JE, Clarke A, Chadwick D, Price DA, Kegg S, Campbell L, Bramham K, Sabin CA, Post FA, Winkler CA; GEN-AFRICA Study Group. GSTM1 Copy Number and Kidney Disease in People With HIV. Kidney Int Rep. 2022 May 13;7(8):1901-1904. doi: 10.1016/j.ekir.2022.05.003. eCollection 2022 Aug. No abstract available. PMID 35967115
- [Background] Hung R, Patel N, Fox J, Cosgrove C, Pett SL, Burns F, Ustianowski A, Rosenvinge M, Bhagani S, Dusheiko G, Childs K, Post FA; GEN-AFRICA study group. Prevalence of HIV/hepatitis B and HIV/hepatitis C coinfection among people of East, South, Central and West African ancestry in the United Kingdom. AIDS. 2021 Aug 1;35(10):1701-1704. doi: 10.1097/QAD.0000000000002929. PMID 33927087
- [Background] Mazaheri T, Buchanan D, Hung R, Campbell L, Hamzah L, Bramham K, Vincent RP, Post FA. Creatinine and cystatin C-based estimated glomerular filtration rate estimates of kidney function in Black people with HIV on antiretroviral therapy. AIDS. 2023 Apr 1;37(5):753-758. doi: 10.1097/QAD.0000000000003466. Epub 2022 Dec 23. PMID 36728909
- [Background] Cechin L, Campbell L, Oliveira A, Goff LM, Post FA. HbA1c screening for diabetes mellitus and to evaluate diabetic control in people of African ancestry with HIV in South London. Int J STD AIDS. 2023 Jun;34(7):484-487. doi: 10.1177/09564624231162163. Epub 2023 Mar 15. PMID 36921326